CLINICAL TRIAL: NCT06200935
Title: Results of the Action of a Combination of Probiotics on the Microbiota and Intestinal Permeability in Children With Neurodevelopmental Disorders and Their Influence on the Improvement of Language, Behavioral Evolution and Learning
Brief Title: Action of Probiotics on the Microbiota and Intestinal Permeability in Children With Neurodevelopmental Disorders and Their Influence on the Improvement of Language and Learning
Status: Completed | Type: Observational
Sponsor: Instituto de Genética Médica y Molecular (Network)
Collaborators: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: MICROBIOTA
Record Dates: First submitted 2023-12-05; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Neurodevelopmental Disorders
Keywords: Neurodevelopment; Probiotics; Microbiota; Learning; Children
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with neurodevelopmental disorders: Boys and girls with neurodevelopmental disorders between 3 and 16 years of age, belonging to two educational centers in Madrid, attended by children with this type of disorders. Both centers have similar characteristics in terms of the type of feeding and management of the children attending them
  Interventions: Dietary Supplement: Probiotic blend

INTERVENTIONS:
Dietary Supplement: Probiotic blend — Administration of one stick of combined probiotics per day for 5 months

SUMMARY:
The study included boys and girls with neurodevelopmental disorders between the ages of 3 and 16 years, belonging to two educational centers in Madrid, attended by children with this type of disorder. Both centers have similar characteristics in terms of the type of feeding and management of the children attending them. The study will be randomized, so that probiotics will be administered to some children and placebos to others; and blinded, so that neither the patient nor his family will know whether probiotic or placebo is administered.

The aim of this project is to study the results obtained on microbiota, intestinal permeability, language, behavior and learning of a probiotic combination that will be administered to children in several educational centers that care for children with neurodevelopmental disorders for 5 months.

DETAILED DESCRIPTION:
The trial was conducted in 4 stages:

* Probiotic development, which will be randomized, so that some children will receive the probiotic and others placebos, and blinded, so that neither the children nor their relatives will know whether they take placebo or probiotic.
* Initial survey to rule out digestive symptoms and resolve possible doubts. Data will be collected on type of housing, location, number of family members, and others. Collection of fecal samples prior to the administration of the probiotic, to carry out a microbiota and intestinal permeability study.
* Administration of the probiotic preparation or placebo to the subjects for 5 months. Monitoring will be done within each center and in the middle of the treatment the doctors will make a face-to-face visit to see the children.
* In the last phase a new online visit is made where a complete clinical history and a survey to rule out digestive symptomatology are evaluated. A neurocognitive evaluation is also done using the SENA behavioral test. New fecal samples are collected for a microbiota and intestinal permeability study following the same procedure as in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Children with neurodevelopmental disorders between 3 and 16 years old
* Similar characteristics in terms of type of food

Exclusion Criteria:

* Digestive symptomatology: gastroesophageal reflux, abdominal pain, flatulence, dysphagia, abdominal distension or constipation

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys and girls with neurodevelopmental disorders between 3 and 16 years of age, belonging to two educational centers in Madrid, which are attended by children with this type of disorders. Both centers have similar characteristics in terms of the type of feeding and management of the children attending them.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Microbiota | Through study completion, an average of 6 months
  Examination of fecal samples
Intestinal permeability | Through study completion, an average of 6 months
  Examination of fecal samples and a complete medical history and a survey aimed mainly at ruling out digestive symptoms

SECONDARY OUTCOMES:
Analyze improvement in language, behavior and learning | Through study completion, an average of 6 months
  By monitoring at the school, asking family members and with a face-to-face visit by the doctor.
  SENA behavioral test is performed at the end of the study
Analyze the outcome in pre-existing digestive disorders | Through study completion, an average of 6 months
  A complete medical history and a survey
Analyze the composition of the microbiota and its improvement | Through study completion, an average of 6 months
  By collecting fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapunzina, Principal Investigator — Instituto de Genética Médica y Molecular (INGEMM)
Locations (1):
- Mencía Hermosa Vicente, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Preparation of a scientific article
Supporting Information: Study Protocol
URL: https://www.fundacionquerer.org/resultado-de-la-accion-de-una-combinacion-de-probioticos/

REFERENCES:
- [Result] Navarro F, Liu Y, Rhoads JM. Can probiotics benefit children with autism spectrum disorders? World J Gastroenterol. 2016 Dec 14;22(46):10093-10102. doi: 10.3748/wjg.v22.i46.10093. PMID 28028357
- [Result] Srikantha P, Mohajeri MH. The Possible Role of the Microbiota-Gut-Brain-Axis in Autism Spectrum Disorder. Int J Mol Sci. 2019 Apr 29;20(9):2115. doi: 10.3390/ijms20092115. PMID 31035684
- [Result] McElhanon BO, McCracken C, Karpen S, Sharp WG. Gastrointestinal symptoms in autism spectrum disorder: a meta-analysis. Pediatrics. 2014 May;133(5):872-83. doi: 10.1542/peds.2013-3995. PMID 24777214
- [Result] Johnson D, Letchumanan V, Thurairajasingam S, Lee LH. A Revolutionizing Approach to Autism Spectrum Disorder Using the Microbiome. Nutrients. 2020 Jul 3;12(7):1983. doi: 10.3390/nu12071983. PMID 32635373
- [Result] Strati F, Cavalieri D, Albanese D, De Felice C, Donati C, Hayek J, Jousson O, Leoncini S, Renzi D, Calabro A, De Filippo C. New evidences on the altered gut microbiota in autism spectrum disorders. Microbiome. 2017 Feb 22;5(1):24. doi: 10.1186/s40168-017-0242-1. PMID 28222761
- [Result] Bezawada N, Phang TH, Hold GL, Hansen R. Autism Spectrum Disorder and the Gut Microbiota in Children: A Systematic Review. Ann Nutr Metab. 2020;76(1):16-29. doi: 10.1159/000505363. Epub 2020 Jan 24. PMID 31982866
- [Result] Liu X, Cao S, Zhang X. Modulation of Gut Microbiota-Brain Axis by Probiotics, Prebiotics, and Diet. J Agric Food Chem. 2015 Sep 16;63(36):7885-95. doi: 10.1021/acs.jafc.5b02404. Epub 2015 Sep 1. PMID 26306709
- [Result] Martin R, Laval L, Chain F, Miquel S, Natividad J, Cherbuy C, Sokol H, Verdu EF, van Hylckama Vlieg J, Bermudez-Humaran LG, Smokvina T, Langella P. Bifidobacterium animalis ssp. lactis CNCM-I2494 Restores Gut Barrier Permeability in Chronically Low-Grade Inflamed Mice. Front Microbiol. 2016 May 6;7:608. doi: 10.3389/fmicb.2016.00608. eCollection 2016. PMID 27199937
- [Result] Hughes KR, Harnisch LC, Alcon-Giner C, Mitra S, Wright CJ, Ketskemety J, van Sinderen D, Watson AJ, Hall LJ. Bifidobacterium breve reduces apoptotic epithelial cell shedding in an exopolysaccharide and MyD88-dependent manner. Open Biol. 2017 Jan;7(1):160155. doi: 10.1098/rsob.160155. PMID 28123052
- [Result] Fornai M, Pellegrini C, Benvenuti L, Tirotta E, Gentile D, Natale G, Ryskalin L, Colucci R, Piccoli E, Ghelardi E, Blandizzi C, Antonioli L. Protective effects of the combination Bifidobacterium longum plus lactoferrin against NSAID-induced enteropathy. Nutrition. 2020 Feb;70:110583. doi: 10.1016/j.nut.2019.110583. Epub 2019 Sep 12. PMID 31739175